CLINICAL TRIAL: NCT05885035
Title: Effects of Calcium Hydroxylapatite on Cellulite Dimples in the Buttocks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kalpna Kay Durairaj, MD, FACS (Other)
Collaborators: Merz North America, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kalpna Kay Durairaj, MD, FACS, Principal Investigator, K. Kay Durairaj, MD, FACS, A Medical Corporation
Organization: K. Kay Durairaj, MD, FACS, A Medical Corporation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD2019
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Cellulite
Keywords: Buttocks; Calcium hydroxylapatite; Hyperdilution; Hyperdiluted calcium hydroxylapatite; Minimally invasive; Gluteal augmentation
MeSH Terms: conditions — Cellulite | interventions — Durapatite

STUDY DESIGN:
Intervention Model Description: The model group will consist of females who present with cellulite dimples in the buttocks. Women are ideal for this study because they have more cellulite dimpling and a predisposition to dimpling due to the anatomy of their fibrous septa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treated with hyperdilute Calcium Hydroxylapatite (CaHA) (Experimental): Subjects will have 3 treatment sessions at weeks 0, 4, and 8 and a final live assessment visit at week 14. Approximately two syringes of CaHA will be injected per side of the buttocks (at sites with cellulite dimpling) during each of the three treatment sessions.
  Interventions: Drug: Calcium Hydroxyapatite

INTERVENTIONS:
Drug: Calcium Hydroxyapatite — Each syringe of CaHA contains 1.5 cc of product, and it will be diluted 1:1 with 1.0 cc of normal saline solution and 0.5 cc of 1% Lidocaine with a ratio of 1:100,000 epinephrine in the target sites.

SUMMARY:
The goal of this clinical trial is to test the efficacy of Calcium Hydroxylapatite (CaHA) in treating cellulite dimples in the buttocks. Participants will:

* have 3 treatment sessions at weeks 0, 4, and 8 and a final live assessment visit at week 14
* receive approximately 2 syringes per side of the buttocks, per treatment session
* have their pictures taken before and after each treatment session, and once more during the final visit

DETAILED DESCRIPTION:
Twenty-five (25) subjects will be enrolled in the study. The patient's body fat composition will be measured by a digital full body composition scale, which will be used to determine the individual percent body fat and eligibility.

The subjects will have three treatment sessions at weeks 0, 4, and 8 and a final live assessment visit at week 14. Office visits will last for approximately two hours. All subjects will have photographs taken before and after each treatment session. Photographs will be taken with buttocks in a relaxed and flexed state. All pictures will be taken via the Quantificare Liveviz Infinity Pro and will be stored via a HIPAA-compliant server.

Subjects will be treated with subdermal injections of CaHA diluted 1:1 with normal saline solution and 1% Lidocaine after having their pictures taken. Subjects will be asked to lay in the prone position with exposed buttocks. Topical Lidocaine/Tetracaine 23%/7% ointment cream will be applied to the treatment sites. After 15 minutes of numbing, the topical anesthetic will be cleaned off with alcohol. Thereafter, subjects will be asked to stand in an upright position to easily mark the areas with cellulite dimpling. The subjects will also be asked to flex and relax their buttocks to let the physician assess the areas of dimpling. Subjects will go back to laying in prone position to receive subdermal injections of CaHA. Multiple, retrograde, linear injections using a standard 25G cannula will be performed with a threading technique by the treating physician. Post injection, a calming cream will be applied to the treated area while massaging in a circular motion for five minutes. Subjects will be called 24-48 hours after each treatment session to check up on comfort and answer questions.

The treating physician will rate each subject's cellulite dimples using the Cellulite Severity Scale (CSS) at each visit. The Global Aesthetic Improvement Scale (GAIS) will be used by the treating physician and subjects to rate aesthetic improvement at each visit after baseline. Subjects will also rate their overall aesthetic improvement and treatment satisfaction at each visit after baseline according to a 5-point scale: (1) Extremely dissatisfied, (2) Dissatisfied, (3) Slightly satisfied, (4) Satisfied, (5) Extremely satisfied. Before and after photos of treated patients will be independently evaluated by the blinded, secondary physician using the CSS scale at each time interval of photos taken.

ELIGIBILITY:
Inclusion Criteria:

* Females, 21-50 years old, of any race and ethnic background.
* 4-5 cellulite dimples that are no deeper than 1 cm each per buttock.
* Body fat between 9% and 55%.
* Written Authorization for Use and Release of Health and Research Study Information has been obtained.
* Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

* Males
* Females who are pregnant, breastfeeding, chronically using nonsteroidal anti-inflammatory drugs, have autoimmune conditions or have a known allergy to the study medications.
* Subjects with piercings or tattoos on the buttocks or those prone to getting keloids.
* Subjects with any aesthetic treatment in the buttocks.
* Subjects with minimal or excessive subcutaneous fat.
* Scars or ongoing infections in the target areas.
* Presence of any clinically significant bleeding disorder or is receiving medication that may increase the risk of bleeding as the result of treatment.
* Subject has a condition or is in a situation which, in the Investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* Any medical condition that would interfere with assessment of safety or efficacy or compromise the subject's ability to undergo study procedures or give informed consent.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 14 weeks
  The treating physician will rate the subject after the final treatment. Based on aesthetic appearance, qualitative success of treatment will be evaluated using the GAIS. Aesthetic appearance will be rated one of the five following options:
  * Worse: The appearance is worse than the original condition
  * No Change: The appearance is essentially the same as the original condition
  * Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated
  * Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result
  * Very Much Improved: Optimal cosmetic result for the treatment in this patient
Cellulite Severity Scale (CSS) Rating | Up to 14 weeks
  The treating physician and the blinded, secondary physician will rate the subject after the final treatment. The scale identifies 5 key clinical morphologic features of cellulite: (1) number of evident depressions, (2) depth of depressions, (3) morphologic appearance of skin surface alterations, (4) grade of laxity, flaccidity, or sagging skin, and (5) the classification scale originally described by Nurnberger and Muller. The scale has 4 points to describe each feature of cellulite: Stage 0 is no dimpling in relaxed or contracted states, Stage 1 implies no dimpling upon relaxed states but dimpling during muscle contraction or skin pinching, Stage 2 implies dimpling appears spontaneously when standing but not when lying down, and Stage 3 implies dimpling is spontaneously present when both standing and lying down and is evident to the naked eye.

SECONDARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 8 weeks
  Based on aesthetic appearance, qualitative success of treatment will be evaluated by the treating physician using the GAIS. Aesthetic appearance will be rated one of the five following options:
  * Worse: The appearance is worse than the original condition
  * No Change: The appearance is essentially the same as the original condition
  * Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated
  * Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result
  * Very Much Improved: Optimal cosmetic result for the treatment in this patient
Global Aesthetic Improvement Scale (GAIS) Rating | Up to 14 weeks
  Based on aesthetic appearance, qualitative success of treatment will be self-evaluated by subjects using the GAIS. Aesthetic appearance will be rated one of the five following options:
  * Worse: The appearance is worse than the original condition
  * No Change: The appearance is essentially the same as the original condition
  * Improved: Obvious improvement in appearance from the initial condition, but a touchup or re-treatment is indicated
  * Much Improved: Marked improvement in appearance but not completely optimal for this patient. A touchup would slightly improve the result
  * Very Much Improved: Optimal cosmetic result for the treatment in this patient
Cellulite Severity Scale (CSS) Rating | Up to 8 weeks
  The treating physician and the blinded, secondary physician will rate the subject at each treatment visit using the CSS Rating. The scale identifies 5 key clinical morphologic features of cellulite: (1) number of evident depressions, (2) depth of depressions, (3) morphologic appearance of skin surface alterations, (4) grade of laxity, flaccidity, or sagging skin, and (5) the classification scale originally described by Nurnberger and Muller. The scale has 4 points to describe each feature of cellulite: Stage 0 is no dimpling in relaxed or contracted states, Stage 1 implies no dimpling upon relaxed states but dimpling during muscle contraction or skin pinching, Stage 2 implies dimpling appears spontaneously when standing but not when lying down, and Stage 3 implies dimpling is spontaneously present when both standing and lying down and is evident to the naked eye.
Patient Satisfaction of Aesthetic Appearance | Up to 14 weeks
  Subjects will rate their satisfaction of aesthetic appearance of their buttocks at each treatment and at the final assessment. Patient satisfaction will be assessed using a 5-point scale: (1) extremely dissatisfied, (2) dissatisfied, (3) slightly satisfied, (4) satisfied, and (5) extremely satisfied.
Patient Treatment Satisfaction | Up to 14 weeks
  Subjects will rate their satisfaction of the treatment at each treatment visit and at the final assessment. Patient satisfaction will be assessed using a 5-point scale: (1) extremely dissatisfied, (2) dissatisfied, (3) slightly satisfied, (4) satisfied, and (5) extremely satisfied.
Telephone Assessment | Up to 14 weeks
  Subjects will be contacted weekly to assess safety injection site and treatment responses. Questionnaire will consist of the 5 following questions:
  1. How are you feeling?
  2. What (if any) side effects are you experiencing?
  3. Are you experiencing pain as a result of treatment?
  4. Are you following the post-procedural instructions?
  5. Do you have any questions or concerns?

CONTACTS AND LOCATIONS:
Overall Officials: Kalpna K Durairaj, MD, Principal Investigator — K. Kay Durairaj, MD, FACS, A Medical Corporation
Locations (1):
- K. Kay Durairaj, MD, FACS, A Medical Corporation, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with interest in calcium hydroxyapatite and cellulite dimpling. Individual participant data that underlies the results reported in this article will be shared after identification. Approval of the request and execution of all applicable agreements (e.g., a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Furthermore, the proposed use of trial IPD must be approved with an Independent Review Committee prior to any data sharing.
Supporting Information: Study Protocol
Time Frame: Data will become available beginning 12 months and ending 28 months after article publication. Upon approval of a data sharing request, data will be accessible to researchers for up to 3 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in scientific research, and will be provided following review and approval of a research proposal, Statistical Analysis Plan (SAP), and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact research@beautybydrkay.com.

REFERENCES:
- [Result] Amore R, Amuso D, Leonardi V, Sbarbati A, Conti G, Albini M, Leva F, Terranova F, Guida A, Gkritzalas K, Gavashely L, Velichenko R. Treatment of Dimpling from Cellulite. Plast Reconstr Surg Glob Open. 2018 May 18;6(5):e1771. doi: 10.1097/GOX.0000000000001771. eCollection 2018 May. PMID 29922557
- [Result] de Almeida AT, Figueredo V, da Cunha ALG, Casabona G, Costa de Faria JR, Alves EV, Sato M, Branco A, Guarnieri C, Palermo E. Consensus Recommendations for the Use of Hyperdiluted Calcium Hydroxyapatite (Radiesse) as a Face and Body Biostimulatory Agent. Plast Reconstr Surg Glob Open. 2019 Mar 14;7(3):e2160. doi: 10.1097/GOX.0000000000002160. eCollection 2019 Mar. PMID 31044123
- [Result] Goldie K, Peeters W, Alghoul M, Butterwick K, Casabona G, Chao YYY, Costa J, Eviatar J, Fabi SG, Lupo M, Sattler G, Waldorf H, Yutskovskaya Y, Lorenc P. Global Consensus Guidelines for the Injection of Diluted and Hyperdiluted Calcium Hydroxylapatite for Skin Tightening. Dermatol Surg. 2018 Nov;44 Suppl 1:S32-S41. doi: 10.1097/DSS.0000000000001685. PMID 30358631
- [Result] Casabona G, Marchese P. Calcium Hydroxylapatite Combined with Microneedling and Ascorbic Acid is Effective for Treating Stretch Marks. Plast Reconstr Surg Glob Open. 2017 Sep 26;5(9):e1474. doi: 10.1097/GOX.0000000000001474. eCollection 2017 Sep. PMID 29062646
- [Result] Loghem JV, Yutskovskaya YA, Philip Werschler W. Calcium hydroxylapatite: over a decade of clinical experience. J Clin Aesthet Dermatol. 2015 Jan;8(1):38-49. PMID 25610523
- [Result] Silvers SL, Eviatar JA, Echavez MI, Pappas AL. Prospective, open-label, 18-month trial of calcium hydroxylapatite (Radiesse) for facial soft-tissue augmentation in patients with human immunodeficiency virus-associated lipoatrophy: one-year durability. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):34S-45S. doi: 10.1097/01.prs.0000234847.36020.52. PMID 16936543
- [Result] Carruthers A, Liebeskind M, Carruthers J, Forster BB. Radiographic and computed tomographic studies of calcium hydroxylapatite for treatment of HIV-associated facial lipoatrophy and correction of nasolabial folds. Dermatol Surg. 2008 Jun;34 Suppl 1:S78-84. doi: 10.1111/j.1524-4725.2008.34247.x. PMID 18547186
- [Result] Goldman MP, Moradi A, Gold MH, Friedmann DP, Alizadeh K, Adelglass JM, Katz BE. Calcium Hydroxylapatite Dermal Filler for Treatment of Dorsal Hand Volume Loss: Results From a 12-Month, Multicenter, Randomized, Blinded Trial. Dermatol Surg. 2018 Jan;44(1):75-83. doi: 10.1097/DSS.0000000000001203. PMID 28562435
- [Result] Breithaupt A, Fitzgerald R. Collagen Stimulators: Poly-L-Lactic Acid and Calcium Hydroxyl Apatite. Facial Plast Surg Clin North Am. 2015 Nov;23(4):459-69. doi: 10.1016/j.fsc.2015.07.007. PMID 26505542
- [Result] Lorenc ZP, Black JM, Cheung JS, Chiu A, Del Campo R, Durkin AJ, Graivier M, Green JB, Kwok GP, Marcus K, Rammos CB, Werschler WP. Skin Tightening With Hyperdilute CaHA: Dilution Practices and Practical Guidance for Clinical Practice. Aesthet Surg J. 2022 Jan 1;42(1):NP29-NP37. doi: 10.1093/asj/sjab269. PMID 34192299
- [Result] Emer J, Sundaram H. Aesthetic applications of calcium hydroxylapatite volumizing filler: an evidence-based review and discussion of current concepts: (part 1 of 2). J Drugs Dermatol. 2013 Dec;12(12):1345-54. PMID 24301235
- [Result] Cogorno Wasylkowski V. Body vectoring technique with Radiesse((R)) for tightening of the abdomen, thighs, and brachial zone. Clin Cosmet Investig Dermatol. 2015 May 19;8:267-73. doi: 10.2147/CCID.S75631. eCollection 2015. PMID 26056483
- [Result] Chao YY, Kim JW, Kim J, Ko H, Goldie K. Hyperdilution of CaHA fillers for the improvement of age and hereditary volume deficits in East Asian patients. Clin Cosmet Investig Dermatol. 2018 Jul 16;11:357-363. doi: 10.2147/CCID.S159752. eCollection 2018. PMID 30038511
- [Result] Jacovella PF. Calcium hydroxylapatite facial filler (Radiesse): indications, technique, and results. Clin Plast Surg. 2006 Oct;33(4):511-23. doi: 10.1016/j.cps.2006.08.002. PMID 17085220
- [Result] Bass LS, Smith S, Busso M, McClaren M. Calcium hydroxylapatite (Radiesse) for treatment of nasolabial folds: long-term safety and efficacy results. Aesthet Surg J. 2010 Mar;30(2):235-8. doi: 10.1177/1090820X10366549. PMID 20442101
- [Result] Kadouch JA. Calcium hydroxylapatite: A review on safety and complications. J Cosmet Dermatol. 2017 Jun;16(2):152-161. doi: 10.1111/jocd.12326. Epub 2017 Mar 1. PMID 28247924
- [Result] Fabi SG, Alhaddad M, Boen M, Goldman M. Prospective Clinical Trial Evaluating the Long-Term Safety and Efficacy of Calcium Hydroxylapatite for Chest Rejuvenation. J Drugs Dermatol. 2021 May 1;20(5):534-537. doi: 10.36849/JDD.5680. PMID 33938688
- [Result] Marmur ES, Phelps R, Goldberg DJ. Clinical, histologic and electron microscopic findings after injection of a calcium hydroxylapatite filler. J Cosmet Laser Ther. 2004 Dec;6(4):223-6. doi: 10.1080/147641704100003048. PMID 16020207
- [Result] Gonzalez N, Goldberg DJ. Evaluating the Effects of Injected Calcium Hydroxylapatite on Changes in Human Skin Elastin and Proteoglycan Formation. Dermatol Surg. 2019 Apr;45(4):547-551. doi: 10.1097/DSS.0000000000001809. PMID 30893178
- [Result] Lapatina NG, Pavlenko T. Diluted Calcium Hydroxylapatite for Skin Tightening of the Upper Arms and Abdomen. J Drugs Dermatol. 2017 Sep 1;16(9):900-906. PMID 28915285
- [Result] Lizzul PF, Narurkar VA. The role of calcium hydroxylapatite (Radiesse) in nonsurgical aesthetic rejuvenation. J Drugs Dermatol. 2010 May;9(5):446-50. PMID 20480786
- [Result] Yutskovskaya YA, Kogan EA. Improved Neocollagenesis and Skin Mechanical Properties After Injection of Diluted Calcium Hydroxylapatite in the Neck and Decolletage:A Pilot Study. J Drugs Dermatol. 2017 Jan 1;16(1):68-74. PMID 28095536
- [Result] Oranges CM, di Summa PG, Giordano S, Kalbermatten DF, Schaefer DJ. A Changing Paradigm: The Brazilian Butt Lift Is Neither Brazilian Nor a Lift-Why It Needs to Be Called Safe Subcutaneous Buttock Augmentation. Plast Reconstr Surg. 2020 Oct;146(4):502e-503e. doi: 10.1097/PRS.0000000000007200. No abstract available. PMID 32639431
- [Result] Casabona G, Pereira G. Microfocused Ultrasound with Visualization and Calcium Hydroxylapatite for Improving Skin Laxity and Cellulite Appearance. Plast Reconstr Surg Glob Open. 2017 Jul 25;5(7):e1388. doi: 10.1097/GOX.0000000000001388. eCollection 2017 Jul. PMID 28831339
- [Result] Hexsel DM, Dal'forno T, Hexsel CL. A validated photonumeric cellulite severity scale. J Eur Acad Dermatol Venereol. 2009 May;23(5):523-8. doi: 10.1111/j.1468-3083.2009.03101.x. Epub 2009 Feb 13. PMID 19220646
- [Derived] Durairaj K, Baker O, Yambao M, Linnemann-Heath J, Shirinyan A. Safety and Efficacy of Diluted Calcium Hydroxylapatite for the Treatment of Cellulite Dimpling on the Buttocks: Results from an Open-Label, Investigator-Initiated, Single-Center, Prospective Clinical Study. Aesthetic Plast Surg. 2024 May;48(9):1797-1806. doi: 10.1007/s00266-023-03815-z. Epub 2024 Jan 22. PMID 38253886